CLINICAL TRIAL: NCT02739828
Title: Post Marketing Observational Study to Assess Quality of Life Changes in Swedish Patients With Moderate or Severe Hidradenitis Suppurativa (HS) After 6 Months on Adalimumab Treatment (HOPE Study)
Brief Title: Post Marketing Observational Study (PMOS) to Assess Quality of Life in Swedish Hidradenitis Suppurativa (HS) Patients
Acronym: HOPE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-692
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2018-05

CONDITIONS: Hidradenitis Suppurativa
Keywords: Quality of life
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Hidradenitis Suppurativa: Patients with moderate or severe HS treated prescribed adalimumab according to the Swedish Summary of Product Characteristics and treated as per routine clinical practice.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Adalimumab
  Other Names: Humira

SUMMARY:
The objective of this study is to assess quality of life (QoL), skin pain, work productivity/activity and health related problems in Swedish patients with moderate to severe HS before and after 6 months treatment with Adalimumab. Participants will be treated in accordance with normal routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hidradenitis Suppurativa
* Prescribed Adalimumab according to the Summary of Product Characteristics (SmPC)
* Willingness to sign and date a Patient Information/Informed Consent Form

Exclusion Criteria:

* Prior biologic treatment discontinued <6 months before the baseline visit
* Patient not able to understand the language of the provided patient questionnaires
* History of non-compliance with medication or a medical history that could enhance non-compliance with medication, as determined by the investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with moderate or severe Hidradenitis Suppurativa
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (11):
- Sweden (11):
  - Universitetssjukhuset Linköping, Linkoping, Västra Götaland County
  - Hallands Hospital Halmstad, Halmstad
  - Blekinge Hospital, Karlskrona
  - Skaraborgs Hospital, Skövde
  - Karolinska Univ Sjukhuset, Solna
  - Kungsholmens Hudklinik, Stockholm
  - Sodersjukhuset, Stockholm
  - Danderyd Hospital, Stockholm
  - Trelleborg Hospital, Trelleborg
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Hidradenitis Suppurativa: Participants with moderate or severe hidradenitis suppurativa (HS) treated prescribed adalimumab according to the Swedish Summary of Product Characteristics and treated as per routine clinical practice.
Period: Overall Study
Arm/Group | Participants With Hidradenitis Suppurativa
Started | 24
Completed | 19
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Groups:
- Participants With Hidradenitis Suppurativa: Participants with moderate or severe HS treated prescribed adalimumab according to the Swedish Summary of Product Characteristics and treated as per routine clinical practice.
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 24
Age, Continuous [Mean (Full Range); unit: years] | 39.5 [21 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 23
  Mixed Race | 1
Dermatology Life Quality Index (DLQI) [Mean (Standard Deviation); unit: units on a scale] — DLQI assesses symptoms and impacts of dermatologic diseases on quality of life. DLQI scores range from 0 to 30, with a higher score indicating a more impaired quality of life.
  units on a scale | 17.1 (7.2)
Participant's Global Assessment of Skin Pain - Numerical Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — The Participant's Global Assessment of Skin Pain NRS was used to assess the worst and average skin pain due to HS. NRS consists of 2 visual analogue scale (VAS) response questions. Skin pain was rated from 0 (no skin pain) to 10 (skin pain as bad as you can imagine) for each.
  units on a scale
    Skin Pain at its Worst | 6.4 (2.95)
    Skin Pain on Average | 4.5 (2.83)
EuroQual 5 Dimensions (EQ-5D) Questionnaire Responses [Count of Participants; unit: Participants] — The EQ-5D is a participant assessment of 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Participants report the extent of their problems with each of the 5 dimensions of health as "some problems/no problems," "some problems/no problems/unable to do," or "none/moderate/extreme."
  Participants
    Mobility: No Problems | 11
    Mobility: Some Problems | 13
    Self-Care: No Problems | 24
    Self-Care: Some Problems | 0
    Usual Activities: No Problems | 10
    Usual Activities: Some Problems | 13
    Usual Activities: Unable to Do | 1
    Pain/Discomfort: None | 0
    Pain/Discomfort: Moderate | 17
    Pain/Discomfort: Extreme | 7
    Anxiety/Depression: None | 7
    Anxiety/Depression: Moderate | 14
    Anxiety/Depression: Extreme | 3
EQ-5D Visual Analogue Scale (VAS) Score [Mean (Standard Deviation); unit: units on a scale] — The EQ-5D VAS records the participant's self-rated health on a scale from 0-100 where increased scores correspond to better health-related quality of life (HRQL). 0 is the 'worst imaginable health state' and 100 is the 'best imaginable health state'. Increased scores correspond to better health state.
  units on a scale | 56.6 (20.98)
Hidradenitis Suppurativa Impact Assessment (HSIA) Overall Score [Mean (Standard Deviation); unit: percent of maximum HS impact] — The HSIA is a disease specific questionnaire measuring the impact the participant experiences associated with HS. HSIA consist of 18 sub-items, 16 of which range from 0 (no impact) to 10 (most negative impact), and 2 items register time at work/school and time away from work/school because of HS. Overall scores are presented as the percent of maximum HS impact (high values indicate a negative HS impact).
  percent of maximum HS impact | 53.9 (24.1)
WPAI-SHP: Work Time Missed Due to Health Problem [Mean (Standard Deviation); unit: percent of work time missed] — The Work Productivity and Activity Impairment-Specific Health Problem (WPAI-SHP) questionnaire is a 6-item questionnaire used to assess work and activity impairment due to symptoms of HS. Work time missed is calculated based on 2 items: (Q2) the number of hours missed from work due to health problems in the past 7 days from visit and (Q4) the number of actual work hours in the past 7 days from visit, using the formula Q2/(Q2+Q4) and converted to percent. Higher numbers indicate greater impairment and less productivity. Population: Participants who were employed at Baseline and had an assessment.
  percent of work time missed
    number analyzed (Participants) | 17
    (all) | 8.5 (25.92)
WPAI-SHP: Impairment While Working Due to Health Problem [Mean (Standard Deviation); unit: percent of impairment while working] — WPAI-SHP is a 6-item participant-assessed questionnaire used to assess work and activity impairment due to symptoms of HS. Calculated based on 1 item: (Q5) to what degree did the disease impair the productivity while working in the past 7 days from visit. The item was measured on a scale from 0 (no effect) to 10 (completely prevented from doing regular activities/ working), using the formula Q5/10 and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity. Population: Participants who were employed at Baseline and had an assessment.
  percent of impairment while working
    number analyzed (Participants) | 16
    (all) | 35 (28.28)
WPAI-SHP: Overall Work Impairment Due to Health Problem [Mean (Standard Deviation); unit: percent of overall work impairment] — WPAI-SHP is a 6-item participant-assessed questionnaire used to assess work and activity impairment due to symptoms of HS. Calculated based on 3 items: (Q2) the number of hours missed from work due to health problems in the past 7 days; (Q4) the number of actual work hours in the past 7 days; and (Q5) to what degree did the disease impair the productivity while working past 7 days, using the formula Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4))x(Q5/10)] and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity. Population: Participants who were employed at Baseline and had an assessment.
  percent of overall work impairment
    number analyzed (Participants) | 16
    (all) | 36.4 (29.59)
WPAI:SHP: Overall Activity Impairment Due to Health Problem [Mean (Standard Deviation); unit: percent of impairment of activity] — WPAI-SHP is a 6-item participant-assessed questionnaire used to assess work and activity impairment due to symptoms of HS. Calculated based on 1 item: (Q6) to what degree did the disease impair the ability to do regular activities in the past 7 days from visit, measured on a scale from 0 (no effect) to 10 (completely prevented from doing regular activities/working), using the formula Q6/10 and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity. Population: Participants who were employed at Baseline and had an assessment.
  percent of impairment of activity
    number analyzed (Participants) | 17
    (all) | 40.6 (32.3)
WPAI:SHP: Overall Activity Impairment Due to Health Problem: Participants Not Employed at Baseline [Mean (Standard Deviation); unit: percent of impairment of activity] — WPAI-SHP is a 6-item participant-assessed questionnaire used to assess work and activity impairment due to symptoms of HS. Calculated based on 1 item: (Q6) to what degree did the disease impair the ability to do regular activities in the past 7 days from visit, measured on a scale from 0 (no effect) to 10 (completely prevented from doing regular activities/working), using the formula Q6/10 and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity. Population: Participants who were not employed at Baseline and had an assessment.
  percent of impairment of activity
    number analyzed (Participants) | 7
    (all) | 51.4 (13.45)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in DLQI at Week 12
Description: DLQI assesses symptoms and impacts of dermatologic diseases on quality of life. DLQI scores range from 0 to 30, with a higher score indicating a more impaired quality of life.
Time Frame: Baseline, Week 12
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants with an assessment at Week 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 18
score on a scale | -7.8 (6.79)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.0001, paired t-test

2. Secondary Outcome: Change From Baseline in DLQI at Week 4
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants with an assessment at Week 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 19
score on a scale | -9.3 (5.94)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p < 0.0001, paired t-test

3. Secondary Outcome: Change From Baseline in DLQI at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants with an assessment at Week 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 18
score on a scale | -9.3 (9.05)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.0004, paired t-test

4. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Skin Pain - NRS at Week 4
Description: The Participant's Global Assessment of Skin Pain NRS was used to assess the worst and average skin pain due to HS. NRS consists of 2 VAS response questions. Skin pain was rated from 0 (no skin pain) to 10 (skin pain as bad as you can imagine) for each.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 19
units on a scale
  Skin Pain at its Worst | -3.2 (3.22)
  Skin Pain on Average | -2.3 (2.45)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Skin pain at its worst. Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.0005, paired t-test
Statistical Analysis 2: Comparison: Participants With Hidradenitis Suppurativa; Skin pain on average. Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.0006, paired t-test

5. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Skin Pain - NRS at Week 12
Description: as for outcome 4
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 18
units on a scale
  Skin Pain at its Worst | -2.9 (2.82)
  Skin Pain on Average | -2.2 (2.46)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0004, paired t-test
Statistical Analysis 2: Comparison: Participants With Hidradenitis Suppurativa; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0016, paired t-test

6. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Skin Pain - NRS at Week 24
Description: as for outcome 4
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 18
units on a scale
  Skin Pain at its Worst | -2.8 (2.66)
  Skin Pain on Average | -1.4 (2.09)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0003, paired t-test
Statistical Analysis 2: Comparison: Participants With Hidradenitis Suppurativa; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0094, paired t-test

7. Secondary Outcome: EQ-5D Questionnaire Responses at Week 4
Description: The EQ-5D is a participant assessment of 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Participants report the extent of their problems with each of the 5 dimensions of health as "some problems/no problems," "some problems/no problems/unable to do," or "none/moderate/extreme."
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 19
Participants
  Mobility: No Problems | 17
  Mobility: Some Problems | 2
  Self-Care: No Problems | 18
  Self-Care: Some Problems | 1
  Usual Activities: No Problems | 16
  Usual Activities: Some Problems | 3
  Usual Activities: Unable to Perform | 0
  Pain/Discomfort: None | 7
  Pain/Discomfort: Moderate | 11
  Pain/Discomfort: Extreme | 1
  Anxiety/Depression: None | 9
  Anxiety/Depression: Moderate | 10
  Anxiety/Depression: Severe | 0

8. Secondary Outcome: EQ-5D Questionnaire Responses at Week 12
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 18
Participants
  Mobility: No Problems | 16
  Mobility: Some Problems | 2
  Self-Care: No Problems | 17
  Self-Care: Some Problems | 1
  Usual Activities: No Problems | 16
  Usual Activities: Some Problems | 2
  Usual Activities: Unable to Perform | 0
  Pain/Discomfort: None | 4
  Pain/Discomfort: Moderate | 13
  Pain/Discomfort: Extreme | 1
  Anxiety/Depression: None | 11
  Anxiety/Depression: Moderate | 7
  Anxiety/Depression: Severe | 0

9. Secondary Outcome: EQ-5D Questionnaire Responses at Week 24
Description: as for outcome 7
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 18
Participants
  Mobility: No Problems | 14
  Mobility: Some Problems | 4
  Self-Care: No Problems | 17
  Self-Care: Some Problems | 1
  Usual Activities: No Problems | 15
  Usual Activities: Some Problems | 2
  Usual Activities: Unable to Perform | 1
  Pain/Discomfort: None | 7
  Pain/Discomfort: Moderate | 10
  Pain/Discomfort: Extreme | 1
  Anxiety/Depression: None | 11
  Anxiety/Depression: Moderate | 6
  Anxiety/Depression: Severe | 1

10. Secondary Outcome: Change From Baseline in EQ-5D VAS Score at Week 4
Description: The EQ-5D VAS records the participant's self-rated health on a scale from 0-100 where increased scores correspond to better HRQL. 0 is the 'worst imaginable health state' and 100 is the 'best imaginable health state'. Change in EQ-5D VAS score was calculated by deducting the final score from the baseline score. Increased scores correspond to better health state.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 19
score on a scale | 9.9 (18.11)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.0278, paired t-test

11. Secondary Outcome: Change From Baseline in EQ-5D VAS Score at Week 12
Description: as for outcome 10
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 18
score on a scale | 11.4 (19.08)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.0215, paired t-test

12. Secondary Outcome: Change From Baseline in EQ-5D VAS Score at Week 24
Description: as for outcome 10
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 18
score on a scale | 8.7 (25.52)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.1652, paired t-test

13. Secondary Outcome: Change From Baseline in HSIA Overall Score at Week 4
Description: The HSIA is a disease specific questionnaire measuring the impact the participant experiences associated with HS. HSIA consist of 18 sub-items, 16 of which range from 0 (no impact) to 10 (most negative impact), and 2 items register time at work/school and time away from work/school because of HS. Overall scores are presented as the percent of maximum HS impact (high values indicate a negative HS impact).
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent of maximum HS impact
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 19
percent of maximum HS impact | -26.7 (23.33)

14. Secondary Outcome: Change From Baseline in HSIA Overall Score at Week 12
Description: as for outcome 13
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of maximum HS impact
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 18
percent of maximum HS impact | -27.1 (20.96)

15. Secondary Outcome: Change From Baseline in HSIA Overall Score at Week 24
Description: as for outcome 13
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent of maximum HS impact
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 18
percent of maximum HS impact | -26 (24.59)

16. Secondary Outcome: WPAI-SHP: Mean Change From Baseline in Work Time Missed Due to Health Problem at Week 4
Description: The 'work time missed due to health problem' was assessed using the WPAI-SHP questionnaire. WPAI-SHP is a 6-item participant-assessed questionnaire used to assess work and activity impairment due to symptoms of HS. The 'work time missed due to health problem' was calculated based on 2 items: (Q2) the number of hours missed from work due to health problems in the past 7 days from visit and (Q4) the number of actual work hours in the past 7 days from visit. The data was calculated using the formula Q2/(Q2+Q4) and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline, Week 4
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants employed at Baseline with a Week 4 assessment.
Measure: Mean (Standard Deviation); unit: percent of work time missed
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 13
percent of work time missed | -6.7 (28.24)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 1.0000, Sign test

17. Secondary Outcome: WPAI-SHP: Mean Change From Baseline in Work Time Missed Due to Health Problem at Week 12
Description: as for outcome 16
Time Frame: Baseline, Week 12
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants employed at Baseline and an assessment at Week 12.
Measure: Mean (Standard Deviation); unit: percent of work time missed
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 10
percent of work time missed | 2 (6.32)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 1.0000, Sign test

18. Secondary Outcome: WPAI-SHP: Mean Change From Baseline in Work Time Missed Due to Health Problem at Week 24
Description: as for outcome 16
Time Frame: Baseline, Week 24
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants employed at Baseline and an assessment at Week 24.
Measure: Mean (Standard Deviation); unit: percent of work time missed
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 11
percent of work time missed | -13.1 (31.75)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.5000, Sign test

19. Secondary Outcome: WPAI-SHP: Mean Change From Baseline in Impairment While Working Due to Health Problem at Week 4
Description: The 'impairment while working due to health problem' was assessed using the WPAI-SHP questionnaire. WPAI-SHP is a 6-item participant-assessed questionnaire used to assess work and activity impairment due to symptoms of HS. The 'impairment while working due to health problem' was calculated based on 1 item: (Q5) to what degree did the disease impair the productivity while working in the past 7 days from visit. The item was measured on a scale from 0 (no effect) to 10 (completely prevented from doing regular activities/working). The data was calculated using the formula Q5/10 and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline, Week 4
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants employed at Baseline with an assessment at Week 4.
Measure: Mean (Standard Deviation); unit: percent of impairment while working
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 12
percent of impairment while working | -17.5 (28)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.1797, Sign test

20. Secondary Outcome: Mean Change From Baseline in Impairment While Working Due to Health Problem at Week 12
Description: as for outcome 19
Time Frame: Baseline, Week 12
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants employed at Baseline with an assessment at Week 12.
Measure: Mean (Standard Deviation); unit: percent of impairment while working
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 10
percent of impairment while working | -15 (24.61)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.4531, Sign test

21. Secondary Outcome: Mean Change From Baseline in Impairment While Working Due to Health Problem at Week 24
Description: as for outcome 19
Time Frame: Baseline, Week 24
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants employed at Baseline with an assessment at Week 24.
Measure: Mean (Standard Deviation); unit: percent of impairment while working
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 10
percent of impairment while working | -14 (16.47)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.0313, Sign test

22. Secondary Outcome: Mean Change From Baseline in Overall Work Impairment Due to Health Problem at Week 4
Description: The 'overall work impairment due to health problem' was assessed using the WPAI-SHP questionnaire. WPAI-SHP is a 6-item participant-assessed questionnaire used to assess work and activity impairment due to symptoms of HS. The 'overall work impairment due to health problem' was calculated based on 3 items: (Q2) the number of hours missed from work due to health problems in the past 7 days from visit; (Q4) the number of actual work hours in the past 7 days from visit; and (Q5) to what degree did the disease impair the productivity while working past 7 days from visit. The data was calculated using the formula Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4))x(Q5/10)] and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline, Week 4
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percent of overall work impairment
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 12
percent of overall work impairment | -17.4 (28.07)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.3438, Sign test

23. Secondary Outcome: Mean Change From Baseline in Overall Work Impairment Due to Health Problem at Week 12
Description: as for outcome 22
Time Frame: Baseline, Week 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percent of overall work impairment
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 10
percent of overall work impairment | -15 (24.61)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.4531, Sign test

24. Secondary Outcome: Mean Change From Baseline in Overall Work Impairment Due to Health Problem at Week 24
Description: as for outcome 22
Time Frame: Baseline, Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: percent of overall work impairment
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 10
percent of overall work impairment | -16.2 (15.85)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.0156, Sign test

25. Secondary Outcome: Mean Change From Baseline in Overall Activity Impairment Due to Health Problem at Week 4
Description: The 'overall activity impairment due to health problem' was assessed using the WPAI-SHP questionnaire. WPAI-SHP is a 6-item participant-assessed questionnaire used to assess work and activity impairment due to symptoms of HS. The 'overall activity impairment due to health problem' was calculated based on 1 item: (Q6) to what degree did the disease impair the ability to do regular activities in the past 7 days from visit. The item was measured on a scale from 0 (no effect) to 10 (completely prevented from doing regular activities/working). The data was calculated using the formula Q6/10 and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline, Week 4
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants employed at Baseline at Week 4.
Measure: Mean (Standard Deviation); unit: percent of impairment of activity
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 14
percent of impairment of activity | -25 (31.32)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.0386, Sign test

26. Secondary Outcome: Mean Change From Baseline in Overall Activity Impairment Due to Health Problem at Week 12
Description: as for outcome 22
Time Frame: Baseline, Week 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percent of impairment of activity
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 13
percent of impairment of activity | -16.2 (29.59)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.3438, Sign test

27. Secondary Outcome: Mean Change From Baseline in Overall Activity Impairment Due to Health Problem at Week 24
Description: as for outcome 22
Time Frame: Baseline, Week 24
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants employed at Baseline assessed at Week 24.
Measure: Mean (Standard Deviation); unit: percent of impairment of activity
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 12
percent of impairment of activity | -15 (42.75)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.1250, Sign test

28. Secondary Outcome: Mean Change From Baseline in Overall Activity Impairment Due to Health Problem at Week 4: Participants Not Employed at Baseline
Description: as for outcome 22
Time Frame: Baseline, Week 4
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants not employed at Baseline with an assessment at Week 4.
Measure: Mean (Standard Deviation); unit: percent of impairment of activity
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 5
percent of impairment of activity | -28 (17.89)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.0625, Sign test

29. Secondary Outcome: Mean Change From Baseline in Overall Activity Impairment Due to Health Problem at Week 12: Participants Not Employed at Baseline
Description: as for outcome 22
Time Frame: Baseline, Week 12
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants not employed at Baseline with an assessment at Week 12.
Measure: Mean (Standard Deviation); unit: percent of impairment of activity
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 5
percent of impairment of activity | -36 (8.94)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.0625, Sign test

30. Secondary Outcome: Mean Change From Baseline in Overall Activity Impairment Due to Health Problem at Week 24: Participants Not Employed at Baseline
Description: as for outcome 22
Time Frame: Baseline, Week 24
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Participants not employed at Baseline with an assessment at Week 24.
Measure: Mean (Standard Deviation); unit: percent of impairment of activity
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 6
percent of impairment of activity | -31.7 (25.63)
Statistical Analysis 1: Comparison: Participants With Hidradenitis Suppurativa; Analysis is under the assumption of completely missing at random (deleted incomplete observations); Test type: Superiority; p = 0.1250, Sign test

31. Secondary Outcome: Percentage of Participants With Hidradenitis Suppurativa Clinical Response (HiSCR) Over Time
Description: HiSCR is a clinical endpoint focusing on assessment of HS inflammatory signs and symptoms to determine the clinical effectiveness of adalimumab.
  HiSCR requires:
  * At least a 50% reduction in the total abscess and inflammatory nodule count (AN count) relative to baseline, and
  * No increase in abscess count, and
  * No increase in draining fistula count. In first bullet AN count is defined as sum of abscess count and inflammatory nodules count.
Time Frame: Week 4, 12 and 24
Population: Full Analysis Set (modified Intention-to-treat): All enrolled participants, with the exception of those who were enrolled and not treated with any dose of adalimumab, or who had no baseline or post baseline data collected for the primary analysis variable DLQI. Observed cases with an assessment at given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With Hidradenitis Suppurativa
Number analyzed (Participants) | 19
percentage of participants
  Week 4 | 73.7 [48.8 to 90.9]
  Week 12: number analyzed (Participants) | 18
  Week 12 | 55.6 [30.8 to 78.5]
  Week 24: number analyzed (Participants) | 18
  Week 24 | 61.1 [35.7 to 82.7]

ADVERSE EVENTS:
Time Frame: Up to 24 Weeks
Arm/Group | Patients With Hidradenitis Suppurativa
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT02739828/SAP_000.pdf
  • Study Protocol (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT02739828/Prot_001.pdf